CLINICAL TRIAL: NCT04482699
Title: Phase I/Phase II Trial of Allogeneic Hybrid TREG/Th2 Cell (RAPA-501-ALLO) Therapy for COVID-19-Related ARDS
Brief Title: RAPA-501-Allo Therapy of COVID-19-ARDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in eligible patient population
Sponsor: Rapa Therapeutics LLC (Industry)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RAPA-501-ALLO-COVID-19
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Severe COVID-19 Disease
Keywords: COVID-19; Allogeneic Hybrid TReg/Th2Cells; RAPA-501-ALLO; Off-the-shelf; Pneumonia; Lung Diseases; Acute Respiratory Distress Syndrome; ARDS; Respiratory Distress Syndrome; 2019 Novel Coronavirus Pneumonia; Acute Lung Injury; Lung Injury; SARS-CoV-2; Cytokine Storm; Corona Virus Infection; Severe Acute Respiratory Syndrome Coronavirus 2; SARS Coronavirus 2; SARS; Reprogram; COVID-19 Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia; Lung Diseases; Respiratory Distress Syndrome; Acute Lung Injury; Lung Injury; Cytokine Release Syndrome; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single agent RAPA-501 cells (dose level 1) (Experimental): Dose level 1 is 40 x 10^6
  Interventions: Biological: RAPA-501-Allo off-the-shelf Therapy of COVID-19
- Single agent RAPA-501 cells (dose level 2) (Experimental): Dose level 2 is 160 x 10^6
  Interventions: Biological: RAPA-501-Allo off-the-shelf Therapy of COVID-19
- RAPA-501 cells (Active Comparator): RAPA-501 cells at either dose level 1 or dose level 2 (whichever has been deemed safe during phase 1)
  Interventions: Biological: RAPA-501-Allo off-the-shelf Therapy of COVID-19
- Placebo-control Cohort (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RAPA-501-Allo off-the-shelf Therapy of COVID-19 — Allogeneic off-the-shelf RAPA-501 cells
  Other Names: RAPA-501-Allo cells
  Arms: RAPA-501 cells; Single agent RAPA-501 cells (dose level 1); Single agent RAPA-501 cells (dose level 2)
Other: Placebo — RAPA-501-Allo cell placebo
  Arms: Placebo-control Cohort

SUMMARY:
The first-in-human Phase 1 study component will evaluate two dose levels of RAPA-501-ALLO off the shelf cells in patients with COVID-19-related ARDS, with key endpoints of safety, biologic and potential disease-modifying effects. The randomized, double-blind, placebo-controlled Phase 2b study component will evaluate infusion of RAPA-501 ALLO off the shelf cells or a control infusion, with the primary endpoint assessing whether RAPA-501 cells reduce 30-day mortality.

The COVID-19 pandemic is a disaster playing out with progressive morbidity and mortality. As of April 6th, 2021, an estimated 132.1 million people have contracted the virus and 2,866,000 deaths have resulted globally. The United States has the highest totals with an estimated 30.8 million people diagnosed and 556,000 deaths. In stages 1 and 2 of COVID-19, viral propagation within the patient is predominant. As such, therapeutic interventions focus on immune molecules (convalescent serum, monoclonal antibodies) and anti-viral medications (remdesivir). In marked contrast, the most severe and deadly form of COVID-19, stage 3, is driven not by viral propagation, but by an out-of-control immune response (hyperinflammation) caused by increases in immune molecules known as cytokines and chemokines. As such, therapeutic interventions for stage 3 disease focus on anti-inflammatory medications such as anti-cytokine therapy (anti-IL-6 drugs) or corticosteroid therapy. Unfortunately, such interventions do not address the full pathogenesis of stage 3 COVID-19, which includes hyperinflammation due to "cytokine storm" and "chemokine storm," tissue damage, hypercoagulation, and multi-organ failure (including lung, heart, kidney and brain). The pulmonary component of stage 3 disease includes acute respiratory distress syndrome (ARDS), which is a final-common-pathway of patient death due to a myriad of conditions, including pneumonia, sepsis, and trauma. There is a dire need for novel cellular treatments that can deliver both a broad-based immune modulation effect and a tissue regenerative effect, such as RAPA-501-ALLO off-the-shelf allogeneic hybrid TREG/Th2 Cells.

Stage 3 COVID-19 carries an estimated 30-day mortality of over 50% in spite of ICU utilization, mechanical ventilation, and supportive care therapies to manage ARDS and multiorgan failure. Narrowly acting targeted anti-inflammatory approaches such as anti-IL-6 therapeutics have not been particularly effective in stage 3 COVID-19 and the broad anti-inflammatory pharmaceutical approach of corticosteroid therapy, has only modestly tempered stage 3 disease in some studies. Cell therapy is also being evaluated in stage 3 COVID-19, in particular, mesenchymal stromal cells (MSC) and now, with the current RAPA-501-ALLO protocol, regulatory T (TREG) cells. TREG therapy has a mechanism of action that includes a multi-faceted anti-inflammatory effect, which puts TREG therapy at the forefront of future curative therapy of a wide range of autoimmune and neurodegenerative diseases, plus transplant complications, such as graft-versus-host disease (GVHD) and graft rejection. In addition, TREG therapy can provide a tissue regenerative effect, which places TREG cell therapy at the lead of novel regenerative medicine efforts to repair a myriad of tissue-based diseases, such as diseases of the skin, muscle, lung, liver, intestine, heart (myocardial infarction) and brain (stroke). RAPA-501-ALLO off-the-shelf cell therapy offers this potential dual threat mechanism of action that incorporates both anti-inflammatory and tissue repair effects for effective treatment of COVID-19 and multiple lethal conditions.

RAPA-501-ALLO cells are generated from healthy volunteers, cryopreserved, banked, and are then available for off-the-shelf therapy anytime. During manufacturing, T cells are "reprogrammed" ex vivo using a novel, patented 7-day two-step process that involves T cell de-differentiation and subsequent re-differentiation towards the two key anti-inflammatory programs, the TREG and Th2 pathways, thus creating a "hybrid" product. The hybrid phenotype inhibits inflammatory pathways operational in COVID-19, including modulation of multiple cytokines and chemokines, which attract inflammatory cells into tissue for initiation of multi-organ damage. The hybrid TREG and Th2 phenotype of RAPA-501-ALLO cells cross-regulates Th1 and Th17 populations that initiate hyperinflammation of COVID-19. RAPA-501 immune modulation occurs in a T cell receptor independent manner, thus permitting off-the-shelf cell therapy. Finally, in experimental models of viral pneumonia and ARDS, TREG cells mediate a protective effect on the lung alveolar tissue. Because of this unique mechanism of action that involves both anti-inflammatory and tissue protective effects, the allogeneic RAPA-501 T cell product is particularly suited for evaluation in the setting of COVID-19-related ARDS.

DETAILED DESCRIPTION:
The first-in-human Phase 1 study component will evaluate two dose levels of RAPA-501-ALLO off the shelf cells in patients with COVID-19-related ARDS, with key endpoints of safety, biologic and potential disease-modifying effects. The randomized, double-blind, placebo-controlled Phase 2b study component will evaluate infusion of RAPA-501 ALLO off the shelf cells or a control infusion, with the primary endpoint assessing whether RAPA-501 cells reduce 30-day mortality.

The COVID-19 pandemic is a disaster playing out with progressive morbidity and mortality. As of April 6th, 2021, an estimated 132.1 million people have contracted the virus and 2,866,000 deaths have resulted globally. The United States has the highest totals with an estimated 30.8 million people diagnosed and 556,000 deaths. The United States has the highest totals with an estimated 22.4 million people diagnosed and 375,000 deaths. In stages 1 and 2 of COVID-19, viral propagation within the patient is predominant. As such, therapeutic interventions focus on immune molecules (convalescent serum, monoclonal antibodies) and anti-viral medications (remdesivir). In marked contrast, the most severe and deadly form of COVID-19, stage 3, is driven not by viral propagation, but by an out-of-control immune response (hyperinflammation) caused by increases in immune molecules known as cytokines and chemokines. As such, therapeutic interventions for stage 3 disease focus on anti-inflammatory medications such as anti-cytokine therapy (anti-IL-6 drugs) or corticosteroid therapy. Unfortunately, such interventions do not address the full pathogenesis of stage 3 COVID-19, which includes hyperinflammation due to "cytokine storm" and "chemokine storm," tissue damage, hypercoagulation, and multi-organ failure (including lung, heart, kidney and brain). The pulmonary component of stage 3 disease includes acute respiratory distress syndrome (ARDS), which is a final-common-pathway of patient death due to a myriad of conditions, including pneumonia, sepsis, and trauma. There is a dire need for novel cellular treatments that can deliver both a broad-based immune modulation effect and a tissue regenerative effect, such as RAPA-501-ALLO off-the-shelf allogeneic hybrid TREG/Th2 Cells.

The mechanism of fatal pneumonia in experimental murine coronavirus infection is mediated by innate inflammasome activation, a resultant robust infiltration of inflammatory monocytes and macrophages, and a subsequent increase in multiple pro-inflammatory cytokines and chemokines. Importantly, the CD4+ and CD8+ adaptive T cell response to experimental coronavirus infection can be either curative or disease propagating. Viral-induced pulmonary inflammation has also been evaluated in non-human primate models, which have confirmed that dysregulated immune activation during viral pneumonia involves T cell subset imbalance, a downstream monocyte-derived inflammatory cascade, and resultant epithelial cell injury. In humans, severity of viral-induced lower respiratory tract infection correlates with increased numbers of effector memory CD8+ T cells in the airway. As recently reviewed, human coronavirus infection represents an ongoing battle between virus and host, with the nature of the response dictating disease cure or alternatively, aggravated lung disease. Evidence exists that the adaptive immune system contributes to pulmonary inflammation during SARS-associated Coronavirus (SARS-CoV) disease: that is, bronchoalveolar fluid from such subjects had increased T cell numbers and increased Th1-associated molecules IL-12, IFN-gamma, and IP-10. This downstream adaptive T cell-mediated inflammatory response is driven in part by the SARS-Co-V protein viroporin 3a. Specifically, viroporin molecules activate the NLRP3 inflammasome that links innate-to-adaptive inflammatory responses. Furthermore, both SARS-CoV and SARS-CoV-2 express an open-reading-frame ORF3a molecule, which also activate the NLRP3 inflammasome.

The nature of immunity during resolution of symptomatic COVID-19 infection has recently been reported, namely: emergence of antibody-secreting cells and CD4+ T follicular helper cells; increase in perforin- and granzyme-expressing CD8+ T cells; and relative lack of an increase in pro-inflammatory cytokines and chemokines. In marked contrast, patients with severe COVID-19 disease had greatly increased plasma levels of cytokines (including IL-2 and TNF-alpha) and chemokines (including IP-10 and MIP-1-alpha) (Huang et al., Lancet, 2020). Collectively, these results indicate that pro-inflammatory cytokine and chemokine responses that occur in severe COVID-19 is detrimental and that effective anti-inflammatory approaches may ultimately prove to be therapeutic. However, as previously detailed, the more advanced Stage 3 COVID-19 disease is characterized by an ARDS component, and cytokine storm, as such, novel approaches to treat the COVID-19 viral pneumonia should optimally incorporate both an anti-inflammatory element and a tissue protection/tissue repair element.

Stage 3 COVID-19 carries an estimated 30-day mortality of over 50% in spite of ICU utilization, mechanical ventilation, and supportive care therapies to manage ARDS and multiorgan failure. Narrowly acting targeted anti-inflammatory approaches such as anti-IL-6 therapeutics have not been particularly effective in stage 3 COVID-19 and the broad anti-inflammatory pharmaceutical approach of corticosteroid therapy, has only modestly tempered stage 3 disease in some studies. Cell therapy is also being evaluated in stage 3 COVID-19, in particular, mesenchymal stromal cells (MSC) and now, with the current RAPA-501-ALLO protocol, regulatory T (TREG) cells. TREG therapy has a mechanism of action that includes a multi-faceted anti-inflammatory effect, which puts TREG therapy at the forefront of future curative therapy of a wide range of autoimmune and neurodegenerative diseases, plus transplant complications, such as graft-versus-host disease (GVHD) and graft rejection. In addition, TREG therapy can provide a tissue regenerative effect, which places TREG cell therapy at the lead of novel regenerative medicine efforts to repair a myriad of tissue-based diseases, such as diseases of the skin, muscle, lung, liver, intestine, heart (myocardial infarction) and brain (stroke). RAPA-501-ALLO off-the-shelf cell therapy offers this potential dual threat mechanism of action that incorporates both anti-inflammatory and tissue repair effects for effective treatment of COVID-19 and multiple lethal conditions.

RAPA-501-ALLO cells are generated from healthy volunteers, cryopreserved, banked, and are then available for off-the-shelf therapy anytime. During manufacturing, T cells are "reprogrammed" ex vivo using a novel, patented 7-day two-step process that involves T cell de-differentiation and subsequent re-differentiation towards the two key anti-inflammatory programs, the TREG and Th2 pathways, thus creating a "hybrid" product. The hybrid phenotype inhibits inflammatory pathways operational in COVID-19, including modulation of multiple cytokines and chemokines, which attract inflammatory cells into tissue for initiation of multi-organ damage. The hybrid TREG and Th2 phenotype of RAPA-501-ALLO cells cross-regulates Th1 and Th17 populations that initiate hyperinflammation of COVID-19. RAPA-501 immune modulation occurs in a T cell receptor independent manner, thus permitting off-the-shelf cell therapy. Finally, in experimental models of viral pneumonia and ARDS, TREG cells mediate a protective effect on the lung alveolar tissue. Because of this unique mechanism of action that involves both anti-inflammatory and tissue protective effects, the allogeneic RAPA-501 T cell product is particularly suited for evaluation in the setting of Stage 3 COVID-19-related ARDS.

In general, classical autoimmune disease, neurodegenerative disease, and viral-induced inflammatory disease are driven by predominance of Th1/Th17-type responses with a relative insufficiency of the counter-regulatory immune suppressive Th2 and TREG subsets. TREG cells, which are defined in part by their expression of FOXP3 transcription factor, have been extensively studied in experimental models for their capacity to modulate autoimmune disease, neurodegenerative disease, and transplantation complications, including graft-versus-host disease (GVHD) and graft rejection. Importantly, T cell production of IL-2 or exogenous IL-2 administration drives lung inflammation during experimental viral infection; therefore, given the known role of TREG cells as a consumer of IL-2, there is a strong mechanistic rationale for a beneficial contribution of TREG cells during viral-driven lung inflammation. Furthermore, in an experimental murine models of virus-induced lung inflammation and lung injury, interventions that augmented TREG cell number and function accelerated the repair of lung injury. And, Th2 cells, which are defined in part by their expression of GATA3 transcription factor, were described thirty years ago as a powerful counter-regulatory population to prevent Th1 cell predominance. It is important to note that clinical data indicates that maneuvers that increase immune suppressive cell populations, including TREG cells, can reduce severe inflammatory disease such as graft-versus-host disease without impairing anti-viral immunity. In addition, in both experimental models and clinical studies, an appropriate level of TREG cells can result in an overall improvement in pulmonary inflammation during viral bronchiolitis. Collectively, these findings indicate that T cells expressing a combined TREG/Th2 phenotype would predictably yield beneficial effects in the setting of viral-induced pulmonary inflammation and injury associated with severe Stage 3 COVID-19 disease.

Clinical trials have evaluated both TREG and Th2-type cells for various conditions, most prominently transplantation complications. In general, thymic-derived natural (n)TREG cells are thought to express a more stable phenotype than post-thymic induced (i)TREG cells; by comparison, iTREG cells can mediate more potent suppression. Nonetheless, both nTREG and iTREG cells are susceptible to differentiation plasticity, which creates concern that a potentially therapeutic TREG population might convert to pathogenic Th1/Th17 phenotypes in vivo. Ex vivo expanded (n)TREG cells were evaluated in the setting of allogeneic hematopoietic cell transplantation (HCT) using cord blood donors; more recently, the same research group has developed ex vivo expanded (i)TREG cell therapy to limit transplant complications. In addition, ex vivo expanded nTREG cells have been evaluated in the setting of type I diabetes mellitus; this clinical trial found that TREG therapy was safe and at least transiently effective in improving disease control. Furthermore, in the setting of amyotrophic lateral sclerosis (ALS), which is a disease propagated by a severe Th1-driven peripheral and central inflammatory response, a clinical trial of nTREG cell adoptive transfer identified that the intervention was safe and showed promise in terms of ALS disease amelioration. Finally, in a phase II study of rapamycin-resistant Th2 cell therapy in the setting of low-intensity allogeneic HCT, adoptive Th2 cell transfer was safe and associated with a shift towards Th2 polarization in vivo, preservation of donor engraftment, stabilization of mixed chimerism, a low rate of GVHD, and potent anti-tumor effects in patients with refractory hematologic malignancy. Collectively, these clinical trial results indicate that the adoptive transfer of TREG and Th2-type populations can be safely administered, even in the allogeneic HCT setting, and can mediate beneficial modulation of inflammatory conditions.

Ex vivo manufacturing can be utilized to generate induced (i)TREG cells from the post-thymic pool of peripheral T cells. In the current protocol, the manufacturing method will focus upon mTOR inhibition, which is an established intervention that promotes the induction of TREG cells. In combination with mTOR inhibition, the culture system that is utilized incorporates cytokines that promote both a Th2 and a TREG phenotype, namely, IL-4, TGF-beta, and IL-2. Finally, the protocol will include a TREG/Th2 cell product comprised of both CD4+ and CD8+ T cell subsets, as these counter-regulatory T cell subsets express differential T cell receptor (TCR) repertoires and a diversity of effector mechanisms that can potentially enhance an anti-inflammatory effect. For RAPA-501 manufacture, peripheral blood mononuclear cells are collected from a steady-state apheresis and subjected to the following two-step culture intervention: in step 1, a severe starvation step results in T cell de-differentiation, which is realized through both selective media utilization and the addition of FDA-approved pharmaceutical agents that potently inhibit mTOR signaling; and in step 2, re-differentiation of T cells occurs using co-stimulation agents and Th2- and TREG-type polarizing cytokines. After 6-days in culture, the resultant TREG/Th2 population is cryopreserved in single-use aliquots at protocol-driven therapeutic doses. T cells of type II cytokine phenotype are characterized in part by their expression of the transcription factor GATA3 whereas regulatory T cell populations are identified in part by their expression of FOXP3 transcription factor. At culture initiation, a very low frequency of T cells express either GATA3 or FOXP3. In contrast, the RAPA-501 cell product manufactured in the TREG/Th2 culture conditions expresses a high frequency of T cells that are either single-positive for GATA3, single-positive for FOXP3, or double-positive for both GATA3 and FOXP3. Importantly, this transcription factor profile is expressed in both manufactured CD4+ and CD8+ T cells. It is important to note that both CD4+ and CD8+ T cell populations with TREG function have been defined, including a CD8+ TREG population that potently suppresses GVHD; it is potentially advantageous to have both subsets represented in a therapeutic product because CD4+ and CD8+ TREG cells utilize differential effector mechanisms.

Regulatory T cell populations can suppress pathogenic effector T cell populations by several defined mechanisms, including through expression of CD39 and CD73 ectonucleotidase molecules, which act to hydrolyse pro-inflammatory ATP towards the immune suppressive adenosine substrate . Indeed, TREG cells that express CD39 possess increased suppressive function and have been associated with resolution of inflammatory bowel disease. Furthermore, suppressive function of human TREG cells is mediated in part by CD73. T cells manufactured in the TREG/Th2 culture condition have an increase in expression of the TREG-associated effector molecules, CD39 and CD73. In addition to the CD39/CD73 ectonucleotidases, TREG cell function has also been correlated with expression of CD103, which is an integrin that dictates epithelial lymphocyte localization. Indeed, CD103 and IL-2 receptor signaling cooperate to maintain immune tolerance in the gut mucosa; furthermore, CD103-expressing TREG cells are critical for amelioration of experimental chronic GVHD . T cells manufactured in the TREG/Th2 culture condition have increased expression of the TREG effector molecule CD103.

In experimental models, the efficacy of adoptive T cell therapy is dependent upon successful engraftment and in vivo T cell persistence. Importantly, the T cell differentiation state helps dictate in vivo persistence, with less differentiated cells having increased persistence. Murine rapamycin-resistant T cells, which expressed a T central memory (TCM) phenotype, had increased in vivo engraftment potential relative to control T cells. In addition, human rapamycin-resistant T cells also had increased engraftment in a human-into-murine model of xenogeneic graft-versus-host disease. T cells with reduced differentiation relative to the T effector memory (TEM) population have increased in vivo persistence and mediate increased in vivo effects, including the TCM subset, the naïve T cell subset, and more recently, the T stem cell memory (TSCM) subset. This relationship between T cell differentiation status and in vivo T cell function is relevant to TREG cells, as: (1) TREG cells of TCM phenotype were more effective at reducing experimental GVHD relative to TREG cells of TEM phenotype; and (2) TREG cells that expressed the stem cell marker CD150 were highly effective for the prevention of stem cell graft rejection. T cells manufactured in the TREG/Th2 culture condition are enriched for cells having a reduced differentiation state consistent with a T stem cell subset, including expression of the CD150 marker.

It is also important to assess the cytokine secretion profile of the manufactured RAPA-501 cells. First, it is critical that the cell product is capable of IL-4 secretion, which is the driver cytokine for subsequent Th2 differentiation. Second, it is desirable that an adoptively transferred T cell population is capable of secreting IL-2, as this capacity indicates a progenitor function that permits T cells to expand more readily in vivo without the need for exogenous IL-2 . Finally, it is important that the RAPA-501 cell population has reduced secretion of the Th1- or Th17-type cytokines IFN-gamma, TNF-alpha, IL-17, and GM-CSF. The manufactured RAPA-501 cell product secretes IL-4 and IL-2 with minimal secretion of Th1- or Th17-type cytokines.

Regulatory T cells can also be defined in part by their ability to suppress the proliferation or function of effector T cells. Importantly, manufactured TREG/Th2 cells potently suppress Th1/Tc1 cell secretion of multiple inflammatory cytokines, including IFN-gamma, GM-CSF, and TNF-alpha. To assess the mechanism of suppression, experiments were performed using the transwell assay, whereby effector T cells and RAPA-501 cells are separated by a filter that prevents cell-to-cell contact but allows cell communication by small soluble mediators such as cytokines. RAPA-501 cells acted in a TCR-independent manner to suppress the cytokine secretion capacity of effector T cells. Because no co-stimulation was provided to the transwell chamber containing RAPA-501 cells, RAPA-501 cells did not require co-stimulation to modulate inflammatory cytokine levels, including IL-2, IFN-gamma, GM-CSF, and TNF-alpha. The following cytokines and chemokines were reduced by RAPA-501 cells in this transwell assay, with relatively equal suppression mediated by CD4+ and CD8+ subsets of RAPA-501 cells: CCL1, CCL2, CCL7, CCL11, CCL13, CCL17, CCL20, CCL22, CCL26, CXCL1, CXCL10, CXCL11, CXCL12, IL-6, IFN-gamma, GM-CSF, and IL-10. The ability of TREG cells to consume IL-2 is a commonly described phenomenon, although previous studies identified the requirement of cell-to-cell contact for IL-2 consumption. As such, RAPA-501 cells are uniquely capable of modulating the level of multiple inflammatory cytokines in a contact-independent manner. These results suggest that RAPA-501 cells represent a suitable candidate for neutralization of multiple cytokines and chemokines associated with various diseases, including viral-induced lung inflammation. In light of this capacity of the RAPA-501 cell product to suppress T cell-mediated inflammation in a TCR-independent manner, RAPA-501 therapy is highly suitable for allogeneic, off-the-shelf treatment applications.

Further experiments were performed to evaluate whether the RAPA-501 cell product might also regulate human CNS microglial cells, which are myeloid-derived cells that are analogous to the peripheral monocyte population. To evaluate whether the RAPA-501 cell product might modulate pro-inflammatory microglial cells in a contact-independent manner, the ability of RAPA-501 cells to reduce the inflammatory state of the microglial cell line HMC3 was tested in a transwell assay. RAPA-501 cells reduced the HMC3 cell secretion of the pro-inflammatory cytokines IL-6 and IFN-gamma and the pro-inflammatory chemokine IP-10 at the relatively low ratio of RAPA-501 cells to microglial cells of 1:40. These results demonstrate that the RAPA-501 product is capable of inhibiting cytokine and chemokine secretion from myeloid-derived populations in a contact- and TCR-independent manner, thereby providing a further rationale for allogeneic, off-the-shelf utilization of the RAPA-501 product.

RAPA-501 cell product for stability of T cell phenotype was also evaluated. That is, it has been determined that a limiting factor of TREG cell therapy may be differentiation plasticity, for example, whereby TREG cells can be influenced by inflammatory cytokines to lose their TREG characteristics and adopt a Th1-type inflammatory state, which may then promote disease pathogenesis. To address this possibility, the RAPA-501 cell capacity to modulate T cell differentiation transcription factors after an extended culture interval that involved T cell co-stimulation, the absence of mTOR inhibitors, and the presence of the polarizing inflammatory cytokines IFN-alpha and IL-6 was studied. These experiments demonstrated that the RAPA-501 cell product had remarkable differentiation stability (continued expression of FOXP3 and GATA3 in CD4+ and CD8+ subsets; lack of up-regulation of TBET).

In summary, RAPA-501 cells express a phenotype consistent with a regulatory T cell population, including: stable expression of the TREG and Th2 transcription factors FOXP3 and GATA3; expression of the TREG functional molecules CD39, CD73, and CD103; expression of a reduced state of T cell differentiation, including expression of the stem cell marker CD150; secretion of a Th2 pattern of cytokines with minimal secretion of Th1/Th17-type cytokines; functional suppressive capacity against both effector Th1/Tc1 cells and pro-inflammatory myeloid cells, including reduced levels of multiple inflammatory cytokines and chemokines; and a capacity to inhibit inflammatory effectors in a contact- and TCR-independent manner. Collectively, these characteristics of the RAPA-501 product predicts that this therapy represents a novel and promising candidate to treat COVID-19-related ARDS.

This is a first-in-human phase 1/phase 2b study evaluating allogeneic RAPA-501 cell therapy in participants with COVID-19-related ARDS. Two phase 1 cohorts will be evaluated, namely, a low-dose Cohort 1 (40 x 10^6 cells/infusion) and a high-dose Cohort 2 (160 x 10^6 cells/infusion); this phase 1 component will utilize dose-limiting-toxicity (DLT) as a primary endpoint. Provided that safety is demonstrated in the phase 1 study component, each RAPA-501 dose cohort can be evaluated in the randomized phase 2b component. In the phase 2b component, for each RAPA-501 dose level determined to be safe, patients will be randomized to receive RAPA-501 cells (n=19) or placebo (n=19). After infusion of either RAPA-501 cells or placebo, these randomized cohorts will continue on standard-of-care therapy (not protocol-driven). The primary endpoint of the phase 2b study is 30-day mortality, with the statistical goal of reducing mortality in RAPA-501 recipients relative to the randomized, placebo-control cohort.

Study participants must be hospitalized patients with COVID-19-related ARDS, specifically: SARS-CoV-2 infection, as determined by RT-PCR or equivalent test; pulmonary infiltrate on radiologic examination; and a diagnosis of ARDS requiring intensive respiratory support including non-invasive ventilation such as high-flow nasal cannula or mechanical ventilation. The study consists of: (1) a study enrollment step (screening); and (2) after eligibility is confirmed, infusion of RAPA-501 cells will be performed. On Cohort 1, infusion of RAPA-501 cells will be at a dose of 40 x 10^6 cells/infusion; three participants will be initially treated, with one week separating participants in this phase 1 component to evaluate for DLT, which will be defined as grade 3 or greater toxicity attributable to RAPA-501 cells within 7-days of infusion. At any point that Cohort 1 therapy is deemed to be safe (either 0/3 or 1/6 having a DLT), then Cohort 1 RAPA-501 therapy can be evaluated in the randomized phase 2b study component to address the primary study objective relating to 30-day mortality. At any point that Cohort 1 therapy is deemed to be safe, treatment on Cohort 2 can be initiated, which will evaluate the infusion of RAPA-501 cells at a dose of 160 x 10^6 cells/infusion. In the same manner as Cohort 1, if Cohort 2 therapy is deemed to be safe, Cohort 2 RAPA-501 therapy can be evaluated in the randomized phase 2b study component to address the primary study objective relating to 30-day mortality. The study will be comprised of three main stages: (1) the above-detailed 30-day interval relating to the primary study objectives; (2) an extended, total 90-day interval to continue relatively intensive clinical monitoring of potential efficacy and safety endpoints; and (3) an extended, total 6-month interval to provide long-term clinical follow-up and to continue to monitor for laboratory parameters relating to immune and viral endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years of age.
2. Participants with SARS-CoV-2 infection, as defined by standard reverse transcriptase polymerase chain reaction (RT-PCR) assay or equivalent test.
3. Must have pulmonary infiltrate on radiologic examination.
4. Participant must have a clinical diagnosis of high-risk ARDS (as defined by a PaO2-to-FiO2 ratio of < 150 mm Hg) requiring intensive respiratory support, including non-invasive methods such as high-flow nasal cannula or mechanical ventilation.
5. AST and ALT ≤ 3 x upper limit of normal (ULN).
6. Consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn at any time without prejudice to future medical care. Informed consent can be obtained from healthcare proxy if the participant is unable to provide consent due to medical status.

Exclusion Criteria:

1. Active uncontrolled infection with a non-COVID-19 agent.
2. Diagnosis of ARDS that is not considered to be high-risk, as defined by PaO2-to-FiO2 ratio of ≥ 150 mm Hg.
3. Any irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%.
4. End-stage liver disease with ascites unrelated to COVID-19 (Childs Pugh score > 12).
5. Uncontrolled or significant cardiovascular disease, including but not limited to: (a) myocardial infarction, stroke, or transient ischemic attack within the past 30 days; (b) uncontrolled angina within the past 30 days; (c) any history of clinically significant arrhythmias such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes; and (d) history of other clinically significant or uncontrolled heart disease, including: cardiomyopathy, congestive heart failure with New York Heart Association functional classification III or IV, myocarditis, pericarditis, or significant pericardial effusion.
6. Known chronic kidney disease of Stage 4 or 5 severity or requiring hemodialysis.
7. COVID-19-associated acute kidney injury requiring dialysis.
8. HIV, hepatitis B, or hepatitis C seropositive.
9. Patients with baseline QTc interval prolongation, as defined by repeated demonstration of a QTc interval >500 milliseconds.
10. Patients on hydroxychloroquine (must discontinue at least 2-days before study entry).
11. Pregnant or breastfeeding participants.
12. Patients of childbearing age, or males who have a partner of childbearing potential, who are unwilling to practice contraception. Effective forms of birth control, which must be continued through the entire on-study 6-month interval, include: Abstinence; Intrauterine device (IUD); Hormonal (birth control pills, injections, or implants); Tubal ligation; or Vasectomy.
13. Participants with malignancy requiring active therapy (not including non-melanoma skin cancer).
14. Recipients of allogeneic hematopoietic cell transplant or solid organ transplant.
15. History of WHO Class III or IV pulmonary hypertension.
16. Severe thromboembolic disease, as defined by: administration of thrombolytic agents, insertion of vena cava filter, or pulmonary thrombectomy within one-week interval prior to screening.
17. Participants may be excluded at the discretion of the PI or if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Through day 7.
  On the phase 1 study component, determine the safety of allogeneic RAPA-501 cells when administered at dose level 1 (Cohort 1, 40 x 106 cells) and dose level 2 (Cohort 2, 160 x 106 cells).
Mortality Rate | 30 days after the first infusion of allogeneic RAPA-501 cells.
  On the phase II study component, determine whether allogeneic RAPA-501 cells result in a mortality rate that is reduced relative to the randomized placebo-control cohort.

SECONDARY OUTCOMES:
Ventilation Support | 90 days after the infusion of allogeneic RAPA-501 cells.
  Number of days requiring intensive respiratory support (either high-flow nasal cannula or mechanical ventilation).
Days of Hospitalization | 90 days after the infusion of allogeneic RAPA-501 cells.
  Number of days of hospitalization among survivors.
Number of Deaths | 90 days after the infusion of allogeneic RAPA-501 cells.
  Number of deaths due to any cause.
Incidence of Infection | 90 days after the infusion of allogeneic RAPA-501 cells.
  Incidence of severe or life-threatening bacterial, invasive fungal, or opportunistic infection.
GVHD Incidence | 90 days after the infusion of allogeneic RAPA-501 cells.
  GVHD incidence and severity.

OTHER OUTCOMES:
Viral Load | Six months after treatment initiation.
  COVID-19 viral load, as determined by standard reverse transcriptase polymerase chain reaction (RT-PCR) assay or equivalent test on nasopharyngeal and/or endotracheal tube swab samples.
Host Immunity | Six months after treatment initiation.
  Development of potentially protective host immunity to COVID-19, as determined by serologic studies.
Peripheral Blood Immune Counts | Six months after treatment initiation.
  Peripheral blood immune counts, including CD4+ and CD8+ T cells, NK cells, and B cells.
T Cell Expression | Six months after treatment initiation.
  T cell expression of co-stimulation molecules (including CD28) and checkpoint receptor molecules (including PD-1).
Peripheral Blood Micro-chimerism | Six months after treatment initiation.
  Peripheral blood micro-chimerism, as determined by PCR amplification of donor and host STR loci.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fowler, M.D., Study Director — Rapa Therapeutics LLC
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No